CLINICAL TRIAL: NCT04569825
Title: Effect of Nasal Steroid in the Treatment of Anosmia Due to COVID-19 Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Anbar (Other)
Responsible Party: Principal Investigator, Raid M. Al-Ani, Proffesor, University Of Anbar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1148
Record Dates: First submitted 2020-09-29; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-08

CONDITIONS: Clinical Trial
Keywords: Anosmia; COVID-19; Nasal steroid
MeSH Terms: conditions — Anosmia; COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Nasal Steroid (Active Comparator): Application of Local Nasal Steroid for the COVID-19 patients with anosmia
  Interventions: Drug: Ophtamesone
- Normal Saline (Placebo Comparator): Application of Normal Saline for the COVID-19 patients with anosmia
  Interventions: Drug: Ophtamesone

INTERVENTIONS:
Drug: Ophtamesone — local application intranasally as drops
  Other Names: Normal Saline

SUMMARY:
Background: Anosmia is a debilitating common symptom of COVID-19. The therapeutic effect of systemic steroid for the treatment of anosmia has been studied with various findings of its efficacy. However, the effect of local steroid was not assessed before.

Objective: To estimate the efficacy of local steroid in the treatment of anosmia in COVID-19 patients.

DETAILED DESCRIPTION:
Background: Anosmia is a debilitating common symptom of COVID-19. The therapeutic effect of systemic steroid for the treatment of anosmia has been studied with various findings of its efficacy. However, the effect of local steroid was not assessed before.

Objective: To estimate the efficacy of local steroid in the treatment of anosmia in COVID-19 patients.

Materials and Methods: A double-blinded randomized controlled trial was conducted at Al-Ramadi Teaching Hospital and Tikrit Teaching Hospital during the period from 23th August to 30th September. Proven cases by real-time polymerase chain reaction and presented with anosmia alone or with ageusia were enrolled in the study. The patients divided into 4 groups according to the treatment modalities. Group A (local steroid nasal drops), group B (local normal saline nasal drops), group C (systemic and local steroid), and group D (systemic steroid and local normal saline). Comparison between the groups concerning the fate and the recovery time of the anosmia was analyzed.

Results and Conclusion: Depends on the finding of the studied patients.

ELIGIBILITY:
Inclusion Criteria: Proven cases of COVID-19 infection by real-time polymerase chain reaction (PCR) of the nasopharyngeal and oropharyngeal swabs and presented with recent onset of anosmia alone or with ageusia or other symptoms of the disease were enrolled in the current study.

-

Exclusion Criteria: Patients with pregnancy, children <18 year, psychological disturbances, previous anosmia, severe sinonasal diseases, previous sinonasal surgery, refuse to participate in the study, and those who lost to follow-up were excluded from the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Recovery rate of anosmia and shorten recovery time | 30 days
  To estimate the recovery rate for both groups and whether nasal steroid enhance the recovery time

CONTACTS AND LOCATIONS:
Overall Officials: Raid M Al-Ani, FIBMS (ENT), Principal Investigator — University Of Anbar
Locations (1):
- Raid Muhmid Al-Ani, Ramadi, Al-Anbar Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Webster KE, O'Byrne L, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the prevention of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD013877. doi: 10.1002/14651858.CD013877.pub3. PMID 36063364
- [Derived] O'Byrne L, Webster KE, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the treatment of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD013876. doi: 10.1002/14651858.CD013876.pub3. PMID 36062970
- [Derived] Rashid RA, Zgair A, Al-Ani RM. Effect of nasal corticosteroid in the treatment of anosmia due to COVID-19: A randomised double-blind placebo-controlled study. Am J Otolaryngol. 2021 Sep-Oct;42(5):103033. doi: 10.1016/j.amjoto.2021.103033. Epub 2021 Apr 7. PMID 33839489